CLINICAL TRIAL: NCT02213289
Title: PANGEA: Personalized Antibodies for Gastro-Esophageal Adenocarcinoma
Brief Title: PANGEA-IMBBP: Personalized Antibodies for Gastro-Esophageal Adenocarcinoma - A 1st Pilot Metastatic Trial of Biologics Beyond Progression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB14-0141
Record Dates: First submitted 2014-08-01; First posted 2014-08-11 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Adenocarcinoma
Keywords: Gastric; Esophagogastric
MeSH Terms: conditions — Adenocarcinoma | interventions — Trastuzumab; depatuxizumab; bemarituzumab; Ramucirumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- ITT-PTS: Personalized Treatment Strategy (Immuno-oncology) (Experimental): For patients with monclonal antibiodies available, initial therapy was tailored based on biomarker profile as follows:
  Immuno-oncology included PD-L1 IHC combined positivity score >10, high microsatellite instability, tumor mutation burden >15 mutations per megabase, and/or Epstein-Barr virus positive. These patients received standard cytotherapy plus Nivolumab.
  Interventions: Drug: Nivolumab; Drug: Standard cytotherapy
- ITT-PTS: Personalized Treatment Strategy (HER2 amplified) (Experimental): HER2 amplified. These patients received standard cytotherapy plus Trastuzumab.
  Interventions: Drug: Trastuzumab; Drug: Standard cytotherapy
- ITT-PTS: Personalized Treatment Strategy (EFGR amplified) (Experimental): EGFR amplified. These patients received ABT-806.
  Interventions: Drug: ABT-806; Drug: Standard cytotherapy
- ITT-PTS: Personalized Treatment Strategy (FGFR2 amplified) (Experimental): FGFR2 amplified. These patients received standard cytotherapy plus Bemarituzumab.
  Interventions: Drug: Bemarituzumab; Drug: Standard cytotherapy
- ITT-PTS: Personalized Treatment Strategy (MAPK/PIK3CA aberrant) (Experimental): MAPK/PIK3CA aberrant. These patients received standard cytotherapy plus Ramucirumab.
  Interventions: Drug: Ramucirumab; Drug: Standard cytotherapy
- ITT-PTS: Personalized Treatment Strategy (EGFR expressing) (Experimental): EGFR expressing. These patients received standard cytotherapy plus ABT 806.
  Interventions: Drug: ABT-806; Drug: Standard cytotherapy
- ITT-PTS: Personalized Treatment Strategy (All negative) (Experimental): All negative. These patients received standard cytotherapy plus Ramucirumab.
  Interventions: Drug: Ramucirumab; Drug: Standard cytotherapy
- Non-ITT: Standard Therapy (Other): Patients without monoclonal antibodies available received standard cytotherapy.
  Interventions: Drug: Standard cytotherapy

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab
  Other Names: Herceptin®
  Arms: ITT-PTS: Personalized Treatment Strategy (HER2 amplified)
Drug: ABT-806 — ABT-806
  Arms: ITT-PTS: Personalized Treatment Strategy (EFGR amplified); ITT-PTS: Personalized Treatment Strategy (EGFR expressing)
Drug: Bemarituzumab — Bemarituzumab
  Arms: ITT-PTS: Personalized Treatment Strategy (FGFR2 amplified)
Drug: Ramucirumab — Ramucirumab
  Other Names: Cyramza
  Arms: ITT-PTS: Personalized Treatment Strategy (All negative); ITT-PTS: Personalized Treatment Strategy (MAPK/PIK3CA aberrant)
Drug: Nivolumab — Nivolumab
  Other Names: Opdivo
  Arms: ITT-PTS: Personalized Treatment Strategy (Immuno-oncology)
Drug: Standard cytotherapy — FOLFOX (First Line) +FOLFIRI (Second Line) +FOLTAX (Third Line)

SUMMARY:
The purpose of this study is to determine if doctors can use the results of special tests of subjects tumor tissue, that will look for specific abnormalities in the tumor, to choose a specific drug that is targeted to work against that abnormality (called molecular profiling) and to see what effects (good and/or bad) that targeted drug has on subjects cancer when it is given with standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic gastric or esophagogastric junction (type I,II,III Siewert) adenocarcinoma
2. Newly-diagnosed chemo-naïve or recurrent after curative-intent surgery

   * >6 months after completion of adjuvant therapy (including chemotherapy and/or radiotherapy)
   * No prior treatment with any targeted agent
   * Patients who have started first line mFOLFOX6 therapy (+/-trastuzumab for HER2 amplified tumors) may be considered for trial participation if they have received no more than 4 doses of therapy at the time of consent and screening.
3. Measurable metastatic disease by RECIST criteria,

   * Must be amenable to ultrasound or CT-guided biopsy of one metastatic lesion
   * Peritoneal disease as the sole site of occult metastasis or presenting as malignant ascites is acceptable if a cell block of tumor cells can be obtained showing >20% viable tumor cells.
4. ECOG PS 0,1
5. Age > 18 years
6. Patients must have normal organ and marrow function as defined below:

   * granulocytes >1,2500/mcL
   * platelets >100,000/mcL
   * total bilirubin < 1.5 x ULN, <1.8 x ULN with liver metastases
   * AST(SGOT)/ALT(SGPT) <2.5 X ULN without liver metastases; <5 X ULN with liver metastases
   * creatinine within normal institutional limits (<1.5) OR
   * creatinine clearance >50 mL/min/1.73m2, (for creatinine level above normal)
   * INR: < 1.5 (patients on warfarin need to be converted to LMWH during study participation to be eligible)
7. Consent to baseline metastatic and progressive disease biopsy (of metastatic/progressing lesion) for enabling biomarker assessment and treatment assignment (at each time point - baseline, PD1, PD2, PD3) as well as for correlative studies.

   • Consent to baseline and serial blood draws for plasma/serum/whole blood banking for correlative studies
8. Ability to understand and the willingness to sign a written informed consent document and consent to the serial nature of the proposed PANGEA treatment with first, second and third line therapy as tolerated.
9. Ability to comply with requirements of the protocol, as assessed by the investigator by the patient signing the consent form.
10. If history of exposure to anthracyclines during perioperative treatment, the following cumulative doses of anthracyclines must be less than:

    Epirubicin < 720 mg/m2 Doxorubicin or liposomal doxorubicin < 360 mg/m2 Mitoxantrone > 120 mg/m2 and idarubicin > 90 mg/m2 If more than one anthracycline has been used, then the cumulative dose must not exceed the equivalent of 360 mg/m2 of doxorubicin.
11. Cardiac Ejection Fraction >50% (for HER2+ patients) as assessed by echocardiogram, MUGA scan, or cardiac MRI
12. Willingness to use effective and reliable methods of contraception (For appropriate methods of contraception considered acceptable see Appendix B).

Both men and women and members of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

1. No CVA within 6 months, no recent MI within 6 months
2. No currently active second malignancy
3. No uncontrolled intercurrent illness or infection
4. No peripheral edema > grade 2 at baseline.
5. No peripheral neuropathy > grade 2 at baseline.
6. No diarrhea > grade 2 at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Catenacci, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ITT-PTS: Personalized Treatment Strategy: For patients with monoclonal antibiodies available, initial therapy was tailored based on biomarker profile as follows:
  Immuno-oncology patients including PD-L1 IHC combined positivity score >10, high microsatellite instability, tumor mutation burden >15 mutations/megabase, and/or Epstein-Barr virus positive received standard cytotherapy plus Nivolumab.
  HER2 amplified patients received standard cytotherapy plus Trastuzumab.
  EGFR amplified patients received standard cytotherapy plus ABT-806
  FGFR2 amplified patients received standard cytotherapy plus Bemarituzumab.
  MAPK/PIK3CA aberrant patients received standard cytotherapy plus Ramucirumab.
  EGFR expressing patients received standard cytotherapy plus ABT 806.
  All negative patients received standard cytotherapy plus Ramucirumab.
  Of note, while the protocol section describes these tailored therapies, the efficacy evaluation was based on pooling these treatments into a combined "personalized treatment strategy" group and comparing with historical controls. Therefore this "arm" includes all such patients with monoclonal antibodies available.
- Non-ITT: Standard Therapy: For patients without monoclonal antibodies available. These patients received standard cytotherapy consisting of FOLFOX (First Line) +FOLFIRI (Second Line) +FOLTAX (Third Line)
  Of note, this arm includes patients without monoclonal antibodies available, for whom no personalized treatment strategy was available. The intent of the protocol was NOT to compare this arm with arm 1.
Period: Overall Study
Arm/Group | ITT-PTS: Personalized Treatment Strategy | Non-ITT: Standard Therapy
Started | 68 | 12
Immuno-oncology | 5 | 0
HER2 Amplified | 16 | 0
EGFR Amplified | 8 | 0
FGFR2 Amplified | 1 | 0
MAPK/PIK3CA Aberrant | 20 | 0
EGFR Expressing | 9 | 0
All Negative | 9 | 0
Other (Non-ITT) | 0 | 12
Completed | 68 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ITT-PTS: Personalized Treatment Strategy: For patients with monclonal antibiodies available, initial therapy was tailored based on biomarker profile as follows:
  Immuno-oncology patients including PD-L1 IHC combined positivity score >10, high microsatellite instability, tumor mutation burden >15 mutations/megabase, and/or Epstein-Barr virus positive patients received standard cytoptherapy plus Nivolumab
  HER2 amplified patients received standard cytotherapy plus Trastuzumab
  EGFR amplified patients received standard cytotherapy plus ABT-806
  FGFR2 amplified patients received standard cytotherapy plus Bemarituzumab
  MAPK/PIK3CA aberrant patients received standard cytotherapy plus Ramucirumab.
  EGFR expressing patients received standard cytotherapy plus ABT 806.
  All negative patients received standard cytotherapy plus Ramucirumab.
- Non-ITT: Standard Therapy: For patients without monoclonal antibodies available, therapy was standard cytotherapy consisting of FOLFOX (First Line) +FOLFIRI (Second Line) +FOLTAX (Third Line)
- Total: Total of all reporting groups
Arm/Group | ITT-PTS: Personalized Treatment Strategy | Non-ITT: Standard Therapy | Total
Number analyzed (Participants) | 68 | 12 | 80
Age, Continuous [Median (Full Range); unit: years] | 61 [28 to 81] | 61 [39 to 77] | 61 [28 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 1 | 16
  Male | 53 | 11 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 0 | 7
  White | 57 | 11 | 68
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 68 | 12 | 80

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Time from enrollment to death from any cause.
Time Frame: Up to 60 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- ITT-PTS: Personalized Treatment Strategy: For patients with monclonal antibiodies available, initial therapy was tailored based on biomarker profile as follows:
  Immuno-oncology patients including PD-L1 IHC combined positivity score >10, high microsatellite instability, tumor mutation burden >15 mutations/megabase, and/or Epstein-Barr virus positive received standard cytotherapy plus Nivolumab.
  HER2 amplified patients received standard cytotherapy plus received Trastuzumab
  EGFR amplified patients received standard cytotherapy plus ABT-806
  FGFR2 amplified patients received standard cytotherapy plus Bemarituzumab.
  MAPK/PIK3CA aberrant patients received standard cytotherapy plus Ramucirumab.
  EGFR expressing patients received standard cytotherapy plus ABT 806.
  All negative patients received standard cytotherapy plus Ramucirumab.
- Non-ITT: Standard Therapy: For patients without monoclonal antibodies available. These patients received standard cytotherapy consisting of FOLFOX (First Line) +FOLFIRI (Second Line) +FOLTAX (Third Line)
Arm/Group | ITT-PTS: Personalized Treatment Strategy | Non-ITT: Standard Therapy
Number analyzed (Participants) | 68 | 12
months | 15.7 [13.4 to 17.7] | 9.0 [4.6 to 20.3]
Statistical Analysis 1: Comparison: ITT-PTS: Personalized Treatment Strategy; Test type: Superiority; p = 0.0024, One-sided Z-test; This was a test of whether the observed 1-year survival rate was significantly different from historical 50% rate

2. Secondary Outcome: Number of Biopsies Leading to an Adverse Event
Description: Number of biopsies leading to an adverse event of the total undergoing baseline biopsies of a primary and metastatic disease site (liver, lung, lymph node, peritoneum/carcinomatosis).
Time Frame: 1 Month
Population: Unit of analysis is the biopsy. Each patient had two biopsies, one of the primary tumor and one of a metastatic site.
Measure: Number; unit: biopsies
Units Other Than Participants: Biopsies
Arm/Group | ITT-PTS: Personalized Treatment Strategy | Non-ITT: Standard Therapy
Number analyzed (Participants) | 68 | 12
Number analyzed (Biopsies) | 136 | 24
biopsies | 1 | 0

3. Secondary Outcome: Completion of Biopsy and Successful, Molecularly-based Treatment Assignment
Description: Completion of biopsies with successful assignment per the treatment algorithm. Biomarker profile assays included next generation sequencing (NGS). EGFR expression was performed by selected-reaction-monitoring mass spectrometry (SRM-MS).
Time Frame: Up to 1 month
Population: Unit of analysis is the biopsy. Two biopsies were performed per patient, one of the primary tumor and one from a metastatic site.
Measure: Number; unit: biopsies
Units Other Than Participants: Biopsies
Arm/Group | ITT-PTS: Personalized Treatment Strategy | Non-ITT: Standard Therapy
Number analyzed (Participants) | 68 | 12
Number analyzed (Biopsies) | 136 | 24
biopsies | 134 | 23

4. Secondary Outcome: Adverse Event From Serial Biopsy for Second-line Treatment
Description: Number of participants with adverse events from serial biopsies of progressing metastatic disease sites (liver, lung, lymph node, peritoneum/carcinomatosis)
Time Frame: Up to 60 Months
Population: This includes subset of patients administered second-line treatment
Measure: Count of Participants; unit: Participants
Arm/Group | ITT-PTS: Personalized Treatment Strategy | Non-ITT: Standard Therapy
Number analyzed (Participants) | 61 | 11
Participants | 0 | 0

5. Secondary Outcome: Completion of Serial Biopsy for Second Line Therapy and Successful, Molecularly-based Treatment Assignment
Description: Completion of biopsy with successful treatment assignment per the treatment algorithm. Biomarker profile assays included next generation sequencing (NGS). EGFR expression was performed by selected-reaction-monitoring mass spectrometry (SRM-MS).
Time Frame: Up to 60 months
Population: This includes subset of patients administered second-line treatment
Measure: Count of Participants; unit: Participants
Arm/Group | ITT-PTS: Personalized Treatment Strategy | Non-ITT: Standard Therapy
Number analyzed (Participants) | 61 | 11
Participants | 51 | 9

6. Secondary Outcome: Adverse Event From Serial Biopsy for Third-line Treatment
Description: as for outcome 4
Time Frame: Up to 60 months
Population: This includes subset of patients administered third-line treatment
Measure: Count of Participants; unit: Participants
Groups:
- ITT-PTS: Personalized Treatment Strategy: For patients with monclonal antibiodies available, initial therapy was tailored based on biomarker profile as follows:
  Immuno-oncology patient including PD-L1 IHC combined positivity score >10, high microsatellite instability, tumor mutation burden >15 mutations/megabase, and/or Epstein-Barr virus positive received standard cytotherapy plus Nivolumab.
  HER2 amplified patients received standard cytotherapy plus received Trastuzumab
  EGFR amplified patients received standard cytotherapy plus ABT-806.
  FGFR2 amplified patients received standard cytotherapy plus Bemarituzumab.
  MAPK/PIK3CA aberrant patients received standard cytotherapy plus Ramucirumab.
  EGFR expressing patients received standard cytotherapy plus ABT 806.
  All negative patients received standard cytotherapy plus Ramucirumab.
Arm/Group | ITT-PTS: Personalized Treatment Strategy | Non-ITT: Standard Therapy
Number analyzed (Participants) | 25 | 3
Participants | 0 | 0

7. Secondary Outcome: Completion of Serial Biopsy for Third Line Therapy and Successful, Molecularly-based Treatment Assignment
Description: as for outcome 5
Time Frame: Up to 60 months
Population: This includes subset of patients administered third-line treatment
Measure: Count of Participants; unit: Participants
Groups:
- ITT-PTS: Personalized Treatment Strategy: For patients with monclonal antibiodies available, initial therapy was tailored based on biomarker profile as follows:
  Immuno-oncology patients including PD-L1 IHC combined positivity score >10, high microsatellite instability, tumor mutation burden >15 mutations/megabase, and/or Epstein-Barr virus positive received standard cytotherapy plus Nivolumab.
  HER2 amplified patients received standard cytotherapy plus received Trastuzumab
  EGFR amplified patients received standard cytotherapy plus ABT-806
  FGFR2 amplified patients received standard cytotherapy plus Bemarituzumab.
  MAPK/PIK3CA aberrant patients received standard cytotherapy plus Ramucirumab.
  EGFR expressing patients received standard cytotherapy plous ABT 806.
  All negative patients received standard cytotherapy plus Ramucirumab.
Arm/Group | ITT-PTS: Personalized Treatment Strategy | Non-ITT: Standard Therapy
Number analyzed (Participants) | 25 | 3
Participants | 21 | 3

8. Other Pre Specified Outcome: First-line Progression-free Survival
Description: Time from enrollment to progression or death during first-line treatment. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 60 Months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- ITT-PTS: Personalized Treatment Strategy: For patients with monclonal antibiodies available, initial therapy was tailored based on biomarker profile as follows:
  Immuno-oncology patients including PD-L1 IHC combined positivity score >10, high microsatellite instability, tumor mutation burden >15 mutations/megabase, and/or Epstein-Barr virus positive received standard cytotherapy plus Nivolumab.
  HER2 amplified patients received standard cytotherapy plus Trastuzumab
  EGFR amplified patients received standard cytotherapy plus ABT-806
  FGFR2 amplified patients received standard cytotherapy plus Bemarituzumab.
  MAPK/PIK3CA aberrant patients received standard cytotherapy plus Ramucirumab.
  EGFR expressing patients received standard cytotherapy plus ABT 806.
  All negative patients received standard cytotherapy plus Ramucirumab.
Arm/Group | ITT-PTS: Personalized Treatment Strategy | Non-ITT: Standard Therapy
Number analyzed (Participants) | 68 | 12
months | 8.2 [7.3 to 9.6] | 6.7 [2.9 to 10.6]

9. Other Pre Specified Outcome: Objective Response to First Line Therapy
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Groups:
- ITT-PTS: Personalized Treatment Strategy: For patients with monclonal antibiodies available, initial therapy was tailored based on biomarker profile as follows:
  Immuno-oncology patients including PD-L1 IHC combined positivity score >10, high microsatellite instability, tumor mutation burden >15 mutations/megabase, and/or Epstein-Barr virus positive received standard cytotherapy plus Nivolumab.
  HER2 amplified patients received standard cytotherapy plus Trastuzumab.
  EGFR amplified patients received standard cytotherapy plus ABT-806.
  FGFR2 amplified patients received standard cytotherapy plus Bemarituzumab.
  MAPK/PIK3CA aberrant patients received standard cytotherapy plus Ramucirumab.
  EGFR expressing patients received standard cytotherapy plus ABT 806.
  All negative patients received standard cytotherapy plus Ramucirumab.
Arm/Group | ITT-PTS: Personalized Treatment Strategy | Non-ITT: Standard Therapy
Number analyzed (Participants) | 54 | 10
Participants | 40 | 4

ADVERSE EVENTS:
Time Frame: 60 months
Description: Molecular arms/groups are combined for this analysis because the intent of the study was to compare the overall strategy of molecular-based treatment vs. not undertaking molecular-based therapy. Thus the number of patients with adverse events over the potential three lines of therapy is reported.
Groups:
- ITT-PTS: Personalized Treatment Strategy: For patients with monclonal antibiodies available, initial therapy was tailored based on biomarker profile as follows:
  Immuno-oncology patients including PD-L1 IHC combined positivity score >10, high microsatellite instability, tumor mutation burden >15 mutations/megabase, and/or Epstein-Barr virus positive received standard cytotherapy plus Nivolumab.
  HER2 amplified patients received standard cytotherapy plus Trastuzumab.
  EGFR amplified patients received standard cytotherapy plus ABT-806..
  FGFR2 amplified patients received standard cytotherapy plus Bemarituzumab.
  MAPK/PIK3CA aberrant patients received standard cytotherapy plus Ramucirumab.
  EGFR expressing patients received standard cytotherapy plus ABT 806.
  All negative patients received standard cytotherapy plus Ramucirumab.
- Non-ITT: Standard Therapy: For patients without monoclonal antibodies available.These patients received standard cytotherapy consisting of FOLFOX (First Line) +FOLFIRI (Second Line) +FOLTAX (Third Line)
Arm/Group | ITT-PTS: Personalized Treatment Strategy | Non-ITT: Standard Therapy
All-Cause Mortality (participants affected / at risk) | 56/68 | 11/12
Serious Adverse Events (participants affected / at risk) | 29/68 | 8/12
Other Adverse Events (participants affected / at risk) | 68/68 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ITT-PTS: Personalized Treatment Strategy (N=68) | Non-ITT: Standard Therapy (N=12)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Death NOS (General disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 4 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Edema limbs (General disorders) | 0 | 1
Esophageal obstruction (Gastrointestinal disorders) | 1 | 0
Esophageal perforation (Gastrointestinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fatigue (General disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Fever (General disorders) | 2 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0
Gastroparesis (Gastrointestinal disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2
Non-cardiac chest pain (General disorders) | 2 | 1
Pelvic infection (Infections and infestations) | 1 | 0
Phlebitis infective (Infections and infestations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Sepsis (Infections and infestations) | 5 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Stroke (Nervous system disorders) | 2 | 0
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ITT-PTS: Personalized Treatment Strategy (N=68) | Non-ITT: Standard Therapy (N=12)
Abdominal distenstion (Gastrointestinal disorders) | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 37 | 7
Alanine aminotransferase increased (Investigations) | 3 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 1
Anemia (Blood and lymphatic system disorders) | 20 | 1
Anorexia (Metabolism and nutrition disorders) | 41 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 8 | 2
Aspartate aminotransferase increased (Investigations) | 4 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 1
Bloating (Gastrointestinal disorders) | 7 | 2
Blood bilirubin increased (Investigations) | 7 | 1
Blurred vision (Eye disorders) | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 2 | 1
Chest pain - cardiac (Congenital, familial and genetic disorders) | 3 | 1
Chills (General disorders) | 6 | 0
Colitis (Gastrointestinal disorders) | 5 | 1
Constipation (Gastrointestinal disorders) | 32 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 5
Diarrhea (Gastrointestinal disorders) | 43 | 5
Dizzines (Nervous system disorders) | 14 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 1
Dysgeusia (Nervous system disorders) | 26 | 4
Dyspepsia/heartburn (Gastrointestinal disorders) | 5 | 1
Dysphagia, esophagitis, odynophagia (Gastrointestinal disorders) | 27 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 | 2
Edema limbs (General disorders) | 20 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 1
Facial pain (Gastrointestinal disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 5 | 2
Fatigue (Gastrointestinal disorders) | 64 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Fever (Gastrointestinal disorders) | 17 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Flu like symptoms (General disorders) | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 1
Gastroesophagial reflux disease (Gastrointestinal disorders) | 13 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 4 | 3
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 1
General disorders and administration site conditions - Other (General disorders) | 6 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 | 1
Hallucinations (Psychiatric disorders) | 0 | 1
Headache (Nervous system disorders) | 10 | 1
Hematuria (Renal and urinary disorders) | 4 | 0
hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 1
Hypertension (Vascular disorders) | 10 | 1
Hypokalemia (Metabolism and nutrition disorders) | 9 | 1
Hypotension (Vascular disorders) | 7 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 8 | 4
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 | 1
Leukocytosis (Cardiac disorders) | 2 | 1
Localized edema (General disorders) | 6 | 1
Mood aleration - depression (Psychiatric disorders) | 10 | 2
Mucositis oral (Gastrointestinal disorders) | 13 | 0
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 52 | 10
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuropathy-sensory (Nervous system disorders) | 58 | 8
Neutrophil count decreased (Investigations) | 8 | 0
Non-cardiac chest pain (General disorders) | 8 | 2
Pain (General disorders) | 20 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 2
Palmar-plantar erythrodysesthesia synrome (Skin and subcutaneous tissue disorders) | 6 | 1
Paresthesia (Nervous system disorders) | 19 | 4
Periodontal disease (Gastrointestinal disorders) | 2 | 1
Platelet count decreases (Investigations) | 14 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Presyncope (Nervous system disorders) | 1 | 1
Proteinuria (Renal and urinary disorders) | 4 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 8 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 1
Renal colic (Renal and urinary disorders) | 1 | 1
Sinusitis (Investigations) | 2 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Thromboembolic event (Vascular disorders) | 9 | 1
Tremor (Nervous system disorders) | 2 | 1
Urinary incontinence (Renal and urinary disorders) | 3 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Upper respiratory infection (Investigations) | 4 | 0
Urinary track infection (Infections and infestations) | 4 | 1
Urinary tract obstruction (Renal and urinary disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 31 | 5
Weight loss (Investigations) | 21 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT02213289/Prot_SAP_000.pdf